CLINICAL TRIAL: NCT04727775
Title: A Retrospective Study of the Effect of Antiviral Drugs on the Treatment of SARS-CoV-2 COVID19
Brief Title: Antiviral Drugs on the Treatment of SARS-CoV-2
Acronym: FavRem
Status: Completed | Type: Observational
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Aidos Konkayev, doctor, Astana Medical University
Other Study IDs: AMU
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Complication of Medical Care; Pneumonia, Viral
MeSH Terms: conditions — Pneumonia, Viral | interventions — favipiravir; remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Complications: Evaluathion
  Interventions: Drug: Favipiravir; Drug: Remdesivir
- Oxygen status: Evaluathion
  Interventions: Drug: Favipiravir; Drug: Remdesivir
- Oxugen support: Evaluathion
  Interventions: Drug: Favipiravir; Drug: Remdesivir

INTERVENTIONS:
Drug: Favipiravir — Antiviral drugs
Drug: Remdesivir — Antiviral drugs

SUMMARY:
Retrospective Non-Randomized Analytical Cohort Study of Completed SARS-CoV2 COVID19 Cases

DETAILED DESCRIPTION:
Analyzing the case histories of patients with SARS-CoV2 COVID19 infection and the impact on the outcomes of prescribing antiviral drugs

ELIGIBILITY:
Inclusion Criteria:

main group

* Patients with COVID19 with medium and easy condition disease
* take favipiravir/remdisivir control group
* Patients with COVID19 with medium and easy condition disease
* not take favipiravir/remdisivir

Exclusion Criteria:

* patients younger 18
* severe conditionis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with previous covid 19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Outcome without comlications | 14 days
  The recovery time will be evaluated with and without antiviral drugs retrospectively in homogeneous groups of patients with SARS-CoV2

SECONDARY OUTCOMES:
Heart rate | 14 days
  Measure
SpO2 | 14 days
  Measure
Blood pressure | 14 days
  Measure
Respiratory rate | 14 days
  Measure

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - Aidos Konkaev, Astana
  - Semey Medical University, Semey

IPD SHARING:
Plan to Share IPD: No
Retrospective study